CLINICAL TRIAL: NCT04698395
Title: Effects of HABIT-ILE in Secondary Brain Damage Outcomes of Infants and Toddlers With Signs of Cerebral Palsy
Brief Title: HABIT-ILE in Infants and Toddlers With Cerebral Palsy (Baby HABIT-ILE)
Acronym: Baby HABIT-ILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University Hospital of Mont-Godinne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B403201316810g
Record Dates: First submitted 2020-12-02; First posted 2021-01-06 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Allocation
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): Baby HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) intervention during two weeks
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)
- Regular care (Active Comparator): Usual customary care intervention during two weeks
  Interventions: Behavioral: Regular care

INTERVENTIONS:
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) — motor learning-based, intensive therapy for children with cerebral palsy
  Other Names: Baby HABIT-ILE
  Arms: HABIT-ILE
Behavioral: Regular care — customary or usual care given to any infant/toddler with cerebral palsy
  Other Names: Usual care
  Arms: Regular care

SUMMARY:
Using a randomized controlled trial design, the possible changes induced by the intensive treatment programme "Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)" in functional, everyday life activities and neuroplastic assessment will be studied in infants and toddlers with cerebral palsy.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, the possible changes in neuroimaging, motor function and everyday life activities of infants and toddlers at risk of or with a diagnosis of cerebral palsy after participating of the intensive treatment programme "Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)" will be studied . Changes, scored by parents in case of questionnaires and by experts in the case of tests, will be observed comparing infants/toddlers after their regular care and after receiving HABIT-ILE. Motor function and daily life activities will be correlated with neuroplastic changes. Moreover, possible therapy onset outcomes differences will be observed.

ELIGIBILITY:
Inclusion Criteria:

* children with diagnosed unilateral cerebral palsy or at risk of developing unilateral cerebral palsy or with signs of unilateral cerebral palsy
* age 8 to 18 months inclusive (corrected age if preterm birth)
* ability to follow instructions and complete testing according to the age.

Exclusion Criteria:

* active seizure
* programmed botulinum toxin or orthopedic surgery in the 6 months previous to the intervention, during intervention period or 6 months after the intervention time.
* severe visual impairments
* severe cognitive impairments
* contraindications to perform magnetic image resonance (MRI) assessments (metal implants, etc.)

Ages: 8 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes on the Mini-Assisting Hand Assessment (Mini-AHA) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Measures how well infants (8-18 months) with signs of unilateral or hemiplegic cerebral palsy use their more affected hand, when using both hands together to play (scored in percentage).

SECONDARY OUTCOMES:
Changes in Bayley Scales of Infant and Toddler Development - Third Edition (BSID-III) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Assess the development of infants and toddlers (1-42 months); three subitems will be considered, the Cognitive Scale, including assessments of attention (familiar and unfamiliar objects, looking for a fallen object, and pretend play), the Language Scale, including understanding and expression of language (recognition of objects and people, following directions, and naming objects and pictures), and the Motor Scale, assessing gross and fine motor skills (including grasping, sitting, stacking blocks, and climbing stairs). Raw scores of the items are converted to scale scores and composite scores (Mean 100, SD 15) ranging from 40 to 160 (higher scores indicates better performance).
Changes in Gross Motor Function Measure - 66 (GMFM-66) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Assess gross motor function of children with cerebral palsy (scored in percentage)
Changes in Visuo-spatial attention assessment with the "Batterie d'évaluation du Jeune Enfant" (BAJE) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Through different simple tasks, measures the visual field, the visuo-motor coordination, the orientation of attention in the space and the eye pursuit.
State of visual impairment of peripheral origin assessed with the standard Battery of Ophthalmological test for infants | baseline
  Clinical assessment will be performed to describe the baseline of the ophthalmological condition. The ophthalmologist search for any abnormal signs of the eyes denoting the presence (or not) of visual impairments.
Changes in Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Parent's filled questionnaire measuring the performance of the child in the daily activities and mobility domains, focusing on the capacity of upper and lower extremities during these activities, computed through the PEDI-CAT software (scores reported in scaled scores).
Changes in Young children's participation and environment measure (YC-PEM) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Based in different children's activities, this parent's filled questionnaire evaluates the level of participation and the quality of the environment in which these activities take place. For each type of activity, caregivers assess 3 dimensions of the child's participation: frequency (8-point scale; 0-7), level of involvement (5-point scale; 1-5), caregiver's percent desire for change (2-points level (y/n) transformed in percentage; 0-100) and perceived impact of environmental support (3-point scale transformed in percentage; 0-100). A software calculates the total score with a maximum of 212
Changes in Canadian Occupational Performance Measure (COPM) | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  In this interview, parents set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the child's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10)
Changes in straightness on kinematics of the upper extremity | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Through a 3D motion system, we measure the percentage of upper extremity trajectory during a reaching task.
Changes in smoothness on kinematics of the upper extremity | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Through a 3D motion system, we measure the variability of the movement during a reaching task.
Changes in time of activity on kinematics of the upper extremity | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Through a 3D motion system, we measure the time from onset to end of the task (in seconds) during a reaching task.
Changes in the quantification of physical activity | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  With a movement sensor on each wrist, the percentage of total time spent in movement (i.e. crawling, walking and running) is measured. Calculated in terms of the changes in the acceleration (m/s2).
Changes in cortical thickness of the brain's gray matter | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Regional brain cortical thickness is acquired from high resolution 3D T1-weighted structural imaging data. For each investigated region, mean cortical metrics (in millimeters) are assessed between the pial surface and the white/grey boundary.
Changes in Fractional Anisotropy (FA) of the corticospinal tract from the motor cortex to the cerebellar peduncle | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  FA is a scalar value (no unit) between 0 and 1 that describes the degree of anisotropy of white matter water molecules. It is measured non-invasively via brain MRI using diffusion tensor imaging (DTI), a modality of Diffusion-Weighted Imaging (DWI). Increased values indicate a higher directionality of the tissue structure.
Changes on the Axial, Radial and Mean Diffusivity (AD, RD, MD) of the corticospinal tract from the motor cortex to the cerebellar peduncle | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  AD, RD and MD are values ranging from 0 to 3.10-3 [mm2/s] that describe the degree of axial, radial and mean molecular diffusion of white matter water molecules. It is measured non-invasively via brain MRI using diffusion tensor imaging (DTI), a modality of Diffusion-Weighted Imaging (DWI). An increased MD can be considered to be an indicator of white matter damage.
Changes on the metrics of the corticospinal tract from the motor cortex to the cerebellar peduncle using the NODDI model | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  The orientation dispersion index (ODI), intracellular volume fraction (ICVF) and the fraction of the isotropic compartment (ISOF) are scalar values ranging from 0 to 1 (no units) that describe the orientation of neural fibers, and the volume fraction of the intracellular and isotropic compartment. It is measured non-invasively via brain MRI using the Neurite Orientation Dispersion and Density Imaging (NODDI) model combined with a Diffusion-Weighted Imaging (DWI) sequence. The results reflects the overall coherence of the fibers, with zero representing highly coherent structures, hence less dispersion of the fibers.
Changes of the fraction and heterogeneity in the neural fibers or isotropic compartments of the corticospinal tract from the motor cortex to the cerebellar peduncle using the DIAMOND model | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  By representing each voxel of the brain as the sum of multiple compartments (representing either a neural fiber population or an isotropic diffusion), the volume fraction ("frac", ranging from 0 to 1, no unit) and heterogeneity ("HEI", ranging from 0 to 1, no unit) of each compartment can be estimated. These metrics are measured non-invasively via brain MRI using the DIstribution of 3D Anisotropic MicrOstructural eNvironments in Diffusion-compartment imaging (DIAMOND) model combined with a Diffusion-Weighted Imaging (DWI) sequence.
Changes in resting-state functional connectivity | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Resting-state functional magnetic resonance imaging (rs-fMRI) evaluates the regional interactions that occur during the resting or task-negative state. The magnitude of the brain activation during rs-fMRI will be assessed
Changes in brain white matter microstructure (WM-μs) using the Microstructure Fingerprinting model | baseline, 3 weeks, 13 weeks and 26 weeks after baseline
  Using a multiple-compartment approach, the signal obtained from a voxel can be estimated as the sum of multiple fiber populations, each presenting a specific fraction ('frac', ranging from 0 to 1, no unit), fiber volume fraction ('fvf', ranging from 0 to 1, no unit) and diffusivity ('diff', in [mm2/s]). On top of those fiber populations, isotropic compartments can also be represented with a specific fraction (frac) and diffusivity (diff). These metrics are measured non-invasively via brain MRI using the Microstructure Fingerprinting model combined with a Diffusion-Weighted Imaging (DWI) sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, PhD, Principal Investigator — MSL-IN Lab, Institute of Neuroscience, UCLouvain; Yves Vandermeeren, MD, PhD, Principal Investigator — Institute of Neuroscience, UCLouvain; CHU-UCL Namur, Neurology Department, UCLouvain
Locations (1):
- Institute of Neuroscience, Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carton de Tournai A, Herman E, Ebner-Karestinos D, Gathy E, Araneda R, Renders A, De Clerck C, Kilcioglu S, Dricot L, Macq B, Vandermeeren Y, Bleyenheuft Y. Hand-Arm Bimanual Intensive Therapy Including Lower Extremities in Infants With Unilateral Cerebral Palsy: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2445133. doi: 10.1001/jamanetworkopen.2024.45133. PMID 39556397
- [Derived] Carton de Tournai A, Herman E, Gathy E, Ebner-Karestinos D, Araneda R, Dricot L, Macq B, Vandermeeren Y, Bleyenheuft Y. Baby HABIT-ILE intervention: study protocol of a randomised controlled trial in infants aged 6-18 months with unilateral cerebral palsy. BMJ Open. 2024 Feb 17;14(2):e078383. doi: 10.1136/bmjopen-2023-078383. PMID 38367973